CLINICAL TRIAL: NCT01559428
Title: The Effects of Plant Sterol and Stanol Esters on Serum Oxyphytosterol Concentrations in Healthy Human Subjects
Brief Title: Phytosterols and Oxyphytosterol Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MEC 09-3-088; TOP grant No. 91208006 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Normocholesterolemic
Keywords: Plant sterols; Plant stanols; Oxyphytosterols; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Plant sterol-enriched margarine (Experimental)
  Interventions: Dietary Supplement: Plant sterol-enriched margarine
- Plant stanol-enriched margarine (Experimental)
  Interventions: Dietary Supplement: Plant stanol-enriched margarine
- Control margarine (Placebo Comparator)
  Interventions: Dietary Supplement: Control margarine

INTERVENTIONS:
Dietary Supplement: Plant sterol-enriched margarine — Daily consumption of 20 gram of a plant sterol-enriched margarine (providing daily 3.0 gram of plant sterols), for a period of 4 weeks. At the end of the 4 weeks, subjects will undergo a postprandial test for 8 hours, in which 20 gram of the plant sterol-enriched margarine is consumed together with a high-fat milkshake
  Arms: Plant sterol-enriched margarine
Dietary Supplement: Plant stanol-enriched margarine — Daily consumption of 20 gram of a plant stanol-enriched margarine (providing daily 3.0 gram of plant stanols), for a period of 4 weeks. At the end of the 4 weeks, subjects will undergo a postprandial test for 8 hours, in which 20 gram of the plant stanol-enriched margarine is consumed together with a high-fat milkshake
  Arms: Plant stanol-enriched margarine
Dietary Supplement: Control margarine — Daily consumption of 20 gram of a control margarine, for a period of 4 weeks. At the end of the 4 weeks, subjects will undergo a postprandial test for 8 hours, in which 20 gram of the control margarine is consumed together with a high-fat milkshake
  Arms: Control margarine

SUMMARY:
Plant sterols and stanols (also called phytosterols and phytostanols) are structurally related to cholesterol, but absorbed to a much lesser extent. Due to this structural similarity, plant sterols and stanols inhibit intestinal cholesterol absorption and lower serum LDL cholesterol concentrations by about 10% at daily intakes of 2.5 g. Plant sterol- and stanol-enriched food products are therefore widely available on the market to lower the risk for coronary heart disease. Plant sterols can undergo oxidation, which results in the formation of oxyphytosterols. Animal studies have now suggested that oxyphytosterols are atherogenic. Although oxyphytosterols have been identified in human serum samples, the effect of an increased intake of plant sterols on serum oxyphytosterol concentrations in humans is not known. On the other hand, plant stanols cannot be oxidized and lower not only cholesterol absorption, but also plant sterol absorption.

The major objective of the present study is to examine the effects of dietary plant sterols and stanols on fasting serum concentrations of oxyphytosterols. The minor objective is to investigate the effects of these products on postprandial serum oxyphytosterol concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 20-30 kg/m2
* mean serum total cholesterol < 7.8 mmol/L
* mean serum triacylglycerol < 3.0 mmol/L
* mean plasma glucose < 6.1 mmol/L

Exclusion Criteria:

* unstable body weight (weight gain or loss > 3 kg in the past two months)
* active cardiovascular diseases like congestive heart failure or recent (<6 months) event (acute myocardial infarction, cerebral vascular incident)
* severe medical conditions that might interfere with the study such as epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel disease and rheumatoid arthritis
* indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus
* use of medication such as corticosteroids, diuretics or lipid lowering therapy
* abuse of drug or alcohol (>21 units per week)
* not willing to stop the consumption of vitamin supplements, fish oil capsules or products rich in sterol or stanol esters 4 weeks before the start of the study (wash-in period)
* use of an investigational product within another biomedical study within the previous month
* pregnant or breast-feeding women
* not willing to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study and during the study
* current smoker
* anemia. with a Hb-level below 7.5 mmol/L for men and below 7.0 mmol/L for women, as indicated by the blood bank of Maastricht

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2010-10-26 (Actual); Study Completion 2012-02-02 (Actual)

PRIMARY OUTCOMES:
Plasma oxyphytosterol concentrations | Measured at baseline and after 4 weeks. Changes will be calculated between day 28 and day 0 of each intervention period.

SECONDARY OUTCOMES:
Serum plant sterol concentrations | Measured at baseline and after 4 weeks. Changes will be calculated between day 28 and day 0 of each intervention period.
Serum lipoprotein concentrations | Measured at baseline and after 3 and 4 weeks. Changes will be calculated between day 21+28 and day 0 of each intervention period.
Plasma glucose concentration | Measured at day 28, on 13 time points
Markers reflecting low-grade inflammation and endothelial activation | Measured at day 28, on 5 time points

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Baumgartner S, Mensink RP, Plat J. Effects of a Plant Sterol or Stanol Enriched Mixed Meal on Postprandial Lipid Metabolism in Healthy Subjects. PLoS One. 2016 Sep 9;11(9):e0160396. doi: 10.1371/journal.pone.0160396. eCollection 2016. PMID 27611192
- [Derived] Baumgartner S, Mensink RP, den Hartog G, Bast A, Bekers O, Husche C, Lutjohann D, Plat J. Oxyphytosterol formation in humans: identification of high vs. low oxidizers. Biochem Pharmacol. 2013 Jul 1;86(1):19-25. doi: 10.1016/j.bcp.2013.02.035. Epub 2013 Mar 13. PMID 23500537
- [Derived] Baumgartner S, Mensink RP, Husche C, Lutjohann D, Plat J. Effects of plant sterol- or stanol-enriched margarine on fasting plasma oxyphytosterol concentrations in healthy subjects. Atherosclerosis. 2013 Apr;227(2):414-9. doi: 10.1016/j.atherosclerosis.2013.01.012. Epub 2013 Jan 21. PMID 23375753
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/23375753
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/23500537
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/25656784
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27611192